CLINICAL TRIAL: NCT05001425
Title: Association Between the Brain Excitability and Postoperative Delirium in Patients Undergoing Heart Valve Replacement Surgery With Cardiopulmonary Bypass: a Prospective Cohort Study
Brief Title: Association Between the Brain Excitability and Postoperative Delirium in Patients Undergoing Heart Valve Replacement Surgery With Cardiopulmonary Bypass
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: LN 2021-1
Record Dates: First submitted 2021-07-27; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Brain Excitability; Postoperative Delirium; Cardiac Surgery
Keywords: Brain excitability; Postoperative Delirium; Abnormal EEG; Excitatory amino acid; Heart valve replacement surgery
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to explorethe brain excitability in patients undergoing heart valve replacement surgery with cardiopulmonary bypass and the correlation with postoperative delirium

DETAILED DESCRIPTION:
Delirium is the most common surgical patients postoperative complications of brain dysfunction. Delirium is a kind of consciousness attention and cognitive function changes of acute brain dysfunction, with volatility and reversibility of postoperative delirium (POD), increased hospital costs and length of hospital stay and mortality rate, and can lower the quality of life, lead to long-term postoperative cognitive dysfunction and dementia. The incidence of postoperative cognitive dysfunction in patients undergoing cardiac valve replacement under cardiopulmonary bypass (CPB) can be as high as 44-53%. However, since the specific mechanism of POD is still not clear, there is still a lack of effective prevention and treatment measures. Therefore, early detection and identification are helpful for the early treatment of POD.When brain injury occurs, the levels of excitatory neurotransmitters (glutamate and aspartate) will rise in a short period of time, and the high concentration of glutamate causes excessive intracellular calcium flow, causing cellular calcium overload, and generating excitatory cytotoxic effects. And abnormal electroencephalogram (EEG) is a kind of due to brain excitability/inhibitory amino acid imbalance caused by brain excitability increased result in abnormal discharge mode, can affect cognitive awareness and activities. Increased brain excitability is harmful to the potential, should avoid to happen. At present, the relationship between brain excitability and POD is still in exploring. Therefore, it is important to clarify the correlation between brain excitability and POD in patients undergoing cardiac valve replacement under CPB for improving the pathogenesis of POD.

ELIGIBILITY:
Inclusion Criteria:

1. ASA Ⅱ - Ⅲ;
2. No cognitive impairment was assessed one day before surgery;
3. Patients undergoing elective heart valve replacement under CPB and signed informed consent.

Exclusion Criteria:

1. Non-CPB surgery, macrovascular surgery, heart transplantation, correction of congenital heart disease;
2. Stroke, schizophrenia, depression, Parkinson's disease, epilepsy or dementia;
3. Inability to communicate with language impairment or major hearing or visual impairment;
4. Liver function child-pugh Grade C, severe liver dysfunction;
5. Severe renal insufficiency requires preoperative renal replacement therapy;
6. A past history of intraoperative knowledge.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients undergoing heart valve replacement surgery with cardiopulmonary bypass
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of delirium after cardiac surgery | The first day after surgery
  Postoperative evaluation delirium occurrence use the The Confusion Assessment Method(CAM) or The Confusion Assessment Method-intensive care unit(CAM-ICU).
The incidence of delirium after cardiac surgery | The second day after surgery
  Postoperative evaluation delirium occurrence use the The Confusion Assessment Method(CAM) or The Confusion Assessment Method-intensive care unit(CAM-ICU).
The incidence of delirium after cardiac surgery | The third day after surgery
  Postoperative evaluation delirium occurrence use the The Confusion Assessment Method(CAM) or The Confusion Assessment Method-intensive care unit(CAM-ICU).
Abnormal EEG during surgery | Complete EEG information from entry to exit of the operating room
  The EEG was collected by Masimo instrument, and the EEG was recognized by the neuroelectrophysiologist, to identify whether the EEG of the patient was epileptic discharge and burst suppression during anesthesia
Plasma excitatory amino acid levels | Before the operation after entering the operating room (baseline)
  Venous blood 5ml was collected and centrifuged (3500r/min,10min)，sera were separated and put into -80 deep temperature refrigerator for testing plasma excitatory amino acid levels.
Plasma excitatory amino acid levels | Immediately after surgery
  Venous blood 5ml was collected and centrifuged (3500r/min,10min)，sera were separated and put into -80 deep temperature refrigerator for testing plasma excitatory amino acid levels.
Plasma excitatory amino acid levels | 24 hours after surgery
  Venous blood 5ml was collected and centrifuged (3500r/min,10min)，sera were separated and put into -80 deep temperature refrigerator for testing plasma excitatory amino acid levels.

CONTACTS AND LOCATIONS:
Overall Officials: Xinli Ni, doctor, Study Chair — General Hospital of Ningxia Medical University
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China